CLINICAL TRIAL: NCT00164879
Title: Endolaparoscopic Versus Immediate Surgery for Obstructing Colorectal Cancers: A Randomised Trial
Brief Title: Endolaparoscopic Versus Immediate Surgery for Obstructing Colorectal Cancers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2002.445-T
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2007-08-07 (Estimated); Status verified 2005-09

CONDITIONS: Colorectal Cancer; Bowel Obstruction
Keywords: Obstructing; Left-sided; Colorectal neoplasms; Obstructing left-sided colorectal cancers
MeSH Terms: conditions — Colorectal Neoplasms; Intestinal Obstruction

INTERVENTIONS:
Procedure: Endoscopic stenting followed by elective laparoscopic resection

SUMMARY:
The aim of this study is to compare the stoma rate, clinical efficacy, and safety of patients treated by endoscopic stenting followed by elective laparoscopic resection (the 'endolaparoscopic approach') versus immediate emergency surgery for obstructing left-sided colorectal cancers.

DETAILED DESCRIPTION:
In patients who present with obstructing left-sided colorectal cancers, emergency surgery carries a significant morbidity and mortality. Traditionally, most of these patients would receive staged operations (Hartmann's procedure). Temporary stoma is often required due to the edematous bowel wall precluding primary anastomosis as a result of obstruction and the poor pre-morbid status. A second operation is subsequently required to restore bowel continuity. Apart from the expensive hospital costs of the staged operations, the patient's acceptance to the stoma is poor and the social inconvenience associated with the stoma is obvious. Thus, a significant portion of patients would not be suitable for the second operation due to poor health or advanced disease and having to bear the stoma for the remainder of life. Recently, self-expandable metal stents have been used with success in relieving the acute obstruction in patients with obstructing left-sided colorectal cancers. Endoscopic stenting may help to relieve the obstruction, avoid emergency surgery, and allows patients to undergo one-stage elective surgery without the necessity of making a stoma. We propose to evaluate the clinical benefits of using self-expandable metal stents in patients with obstructing left-sided colorectal cancers followed by elective laparoscopic resection and compare its use to immediate emergency surgery.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with obstructing colorectal cancers, confirmed on water-soluble contrast enema or computed tomography (CT) scan
* Consented patients

Exclusion Criteria:

* Patients with peritonitis that required immediate surgical intervention
* Patients with distal rectal cancers that are not suitable for stenting
* Moribund patients, unfit for surgery otherwise
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2000-01

PRIMARY OUTCOMES:
The success rate of relieving obstruction after stent insertion
The stoma rate in the two groups of patients

SECONDARY OUTCOMES:
Morbidity and mortality rates in the two groups
Hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: James YW Lau, MD, FRCS(Edin), Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Centre, Prince of Wales Hospital, Hong Kong SAR, China